CLINICAL TRIAL: NCT06774859
Title: A Phase III, Randomized, Open-Label, Active-Controlled Study to Assess the Safety, Pharmacokinetics, and Efficacy of Baloxavir Marboxil in Chinese Pediatric Patients 1 to <12 Years of Age With Influenza Symptoms
Brief Title: Study to Assess the Safety, Pharmacokinetics, and Efficacy of Baloxavir Marboxil in Chinese Pediatric Participants 1 to <12 Years of Age With Influenza Symptoms
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YV44465
Record Dates: First submitted 2025-01-09; First posted 2025-01-14 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human | interventions — baloxavir; Oseltamivir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Baloxavir Marboxil (Experimental): Participants will receive a single oral dose of baloxavir marboxil on Day 1 based on body weight.
  Interventions: Drug: Baloxavir Marboxil
- Oseltamivir (Active Comparator): Participants will receive oseltamivir twice a day for 5 days based on body weight.
  Interventions: Drug: Oseltamivir

INTERVENTIONS:
Drug: Baloxavir Marboxil — Baloxavir marboxil will be administered as oral suspension: 2 milligrams per kilograms (mg/kg) (if weight < 20 kg), 40 mg (if weight ≥ 20 kg to < 80 kg), or 80 mg (if weight ≥ 80 kg).
  Arms: Baloxavir Marboxil
Drug: Oseltamivir — Oseltamivir will be administered as oral capsule: 30 mg (if weight ≤15 kg), 45 mg (if weight > 15 kg to ≥ 23 kg), 60 mg (if weight > 23 kg to ≤ 40 kg) or 75 mg (if weight > 40 kg), twice daily (BID) for 5 days.
  Arms: Oseltamivir

SUMMARY:
The purpose of this study is to evaluate the safety of a single dose baloxavir marboxil compared with 5 days of oseltamivir administered twice a day (BID) in Chinese pediatric participants aged 1 to < 12 years with influenza symptoms.

ELIGIBILITY:
Inclusion Criteria:

* A participant who has a diagnosis of influenza virus infection and meets all the following conditions:

  * Fever ≥ 38°C (tympanic temperature) at screening
  * At least one of the respiratory symptoms of influenza virus infection
* A rapid influenza diagnostic test (RIDT) or polymerase chain reaction (PCR) shows positive for influenza A/B, e.g., point-of-care/local laboratory results with use of nasal aspirate, throat swab, or nasal drip/droplet (or other appropriate sample)
* The time interval between the onset of symptoms and screening is ≤ 48 hours
* PCR (-) or antigen test (-) for severe acute respiratory virus-coronavirus 2 (SARS-CoV-2) using point-of-care/local laboratory test with nasal aspirate, throat swab, or nasal drip/droplet (or other appropriate sample)

Exclusion Criteria:

* A participant having severe influenza virus infection symptoms requiring inpatient treatment
* Received systemic corticosteroid or immunosuppressive therapy
* Primary immunodeficiency syndrome
* History of organ transplantation
* Human immunodeficiency virus (HIV) infection
* Immunization with a live/attenuated influenza vaccine in 2 weeks prior to randomization
* Previous malignancy within the last 5 years or has an active cancer at any site
* A participant who received any medications with anti-flu effect such as baloxavir, peramivir, oseltamivir, zanamivir, favipiravir, arbidol, amantadine or traditional Chinese anti-influenza medicines within 30 days before screening
* Diagnosed with or suspected SARS-CoV-2 infection, or close contacts of diagnosed or suspected SARS-CoV-2 infected patients
* Severe underlying disease or condition potentially affecting study evaluation in the opinion of the investigator/sub-investigator
* A participant who received an investigational or unapproved drug product within 30 days or 5 x the half-life before screening, whichever is longer

Ages: 1 Year to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2024-10-27 (Actual); Primary Completion 2025-05-08 (Actual); Study Completion 2025-05-08 (Actual)

PRIMARY OUTCOMES:
Number of Adverse Events (AEs) and Serious Adverse Events (SAEs) | Up to Day 29

SECONDARY OUTCOMES:
Time to Alleviation of Influenza Signs and Symptoms | Up to Day 15
  Time to Alleviation of Influenza Signs & Symptoms is defined as length of time taken from the start of treatment to the point at which all of the following criteria are met & remain so, for at least 21.5 hours: Score of 0 (no problem) or 1 (minor problem) for cough & nasal symptoms (Items 14 &15 of the Canadian Acute Respiratory Illness & Flu Scale [CARIFS]); "Yes" response to the following question on CARIFS: "Since the last assessment has the subject been able to return to day care/school (if applicable), or resume his or her normal daily activity in the same way as performed prior to developing the flu?" (if possible) & return to afebrile state (tympanic temperature ≤ 37.2°C.
Duration of Fever | Up to Day 15
  Length of time taken by participants to return to afebrile state (tympanic temperature ≤ 37.2°C) and remaining so, for at least 21.5 hours.
Duration of Symptoms | Up to Day 15
  Duration of symptoms is alleviation of all symptoms as defined by a score of 0 [no problem] or 1 [minor problem] and remaining so, for at least 21.5 hours, for all 18 symptoms specified in the CARIFS questionnaire.
Time to Return to Normal Health and Activity Based on the CARIFS Questionnaire | Up to Day 15
  CARIFS parental questionnaire is composed of 18 questions, each with a 4-point ordinal scale (no problem=0 to major problem=3) to measure the duration of illness. Total score ranges from 0 (best possible health) to 54 (worst possible health).
Frequency of Influenza-Related Complications | Up to Day 29
  Influenza related complications include death, hospitalization, radiologically confirmed pneumonia, bronchitis, sinusitis, otitis media, encephalitis/encephalopathy, febrile seizures, myositis.
Percentage of Participants Requiring Antibiotics for Influenza Related Complications | Up to Day 29
Time to Cessation of Viral Shedding as Assessed by Virus Titer | Day 1 to Day 29
Time to Cessation of Viral Shedding as Assessed by Reverse Transcriptase-Polymerase Chain Reaction (RT-PCR) | Day 1 to Day 29
Change From Baseline in Influenza Virus Titer | Baseline (Day 1), Day 2, 4, 6, 10, 15 and 29
Change From Baseline in the Amount of Virus RNA (Based on RT-PCR) | Baseline (Day 1), Day 2, 4, 6, 10, 15 and 29
Percentage of Participants With Positive Influenza Virus Titer | Day 2, 4, 6, 10, 15 and 29
Percentage of Participants With Positive for Influenza Virus as Assessed by RT-PCR | Day 2, 4, 6, 10, 15 and 29
Area Under the Curve (AUC) in Virus Titer | Day 1 to Day 29
Area Under the Curve in Amount of Virus RNA (Based on RT-PCR) | Day 1 to Day 29
Plasma Concentrations of S-033447 | Up to 72 hours post dose
  S-033447 is an active metabolite of baloxavir marboxil.
Area Under the Concentration-time Curve Extrapolated to Infinity (AUCinf) of S-033447 | Up to Day 10
  S-033447 is an active metabolite of baloxavir marboxil.
Maximum Observed Concentration (Cmax) of S-033447 | Up to Day 10
  S-033447 is an active metabolite of baloxavir marboxil.
Time of Maximum Observed Concentration (Tmax) of S-033447 | Up to Day 10
  S-033447 is an active metabolite of baloxavir marboxil.
Elimination Half-life (t1/2) of S-033447 | Up to Day 10
  S-033447 is an active metabolite of baloxavir marboxil.
Polymorphic and Treatment-emergent Amino Acid Substitutions in the PA Gene | Baseline (Day 1) up to Day 29
  Sanger sequencing of the influenza PA gene will be performed to evaluate the incidence of polymorphic (baseline vs. reference) and treatment-emergent (post-baseline vs. baseline) amino acid substitutions.
Effective Concentration (EC50) of Baloxavir Marboxil Evaluated by ViroSpot™ Assay | Up to Day 29
Percentage of Participants with Responses to Palatability and Acceptability Questionnaire | Day 1
  A two-question palatability and acceptability questionnaire will be used. The palatability question ask the participant about taste of the medicine with responses from 'Like very much' to 'Dislike Very Much'. The acceptability question asks participants if they would be happy to take the medicine again, with responses as 'Yes', 'No' and 'Not Sure'.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (18):
- China (18):
  - The First People's Hospital of Changde, Changde
  - Peoples Hospital of Hunan Province, Changsha
  - Hunan Provincial Maternal and Child Health Care Hospital, Changsha
  - Chengdu Women's and Children's Central Hospital, Chengdu
  - Chongqing University Jiangjin Hospital, Chongqing
  - Childern's Hospital of Chongqing Medical University, Chongqing
  - Cnpc Central Hospital, Langfang
  - Liaocheng people's Hospital, Liaocheng
  - Linfen Central Hospital, Linfen
  - Liuzhou People's Hospital, Liuchow
  - Ningbo Women and Children's Hospital, Ningbo
  - Sanmenxia Central Hospital, Sanmenxia
  - The Third People's Hospital of Hainan Province, Sanya
  - The Second Affiliated Hospital of Shantou University Medical College, Shantou
  - The First Affiliated Hospital, Shaoyang University, Shaoyang
  - University of Chinese Academy of Sciences Shenzhen Hospital, Shenzhen
  - Xiamen Maternal and Child Health Hospital, Xiamen
  - Yuncheng Central Hospital, Yuncheng

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing